CLINICAL TRIAL: NCT01076309
Title: Corneal Endothelium Cell Loss After Cataract Extraction in Patients Taking Systemic Sympathetic Alfa-1-a-antagonist Medication (Tamsulosin)
Brief Title: Corneal Endothelium Cell Loss After Cataract Extraction in Patients Taking Tamsulosin
Status: Completed | Type: Observational
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Allan Storr-Paulsen, Frederiksberg University Hospital
Other Study IDs: FH4
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-01

CONDITIONS: Cataract
Keywords: cataract surgery; tamsulosin; endothelium cell
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tamsulosin: Patients taking tamsulosin
- Non-tamsulosin: Patients not taking tamsulosin.

SUMMARY:
The purpose of this study is to determine whether corneal endothelium cell loss during cataract surgery is higher in patients taking Tamsulosin.

DETAILED DESCRIPTION:
Cataract surgery in patients taking Tamsulosin is regarded as more challenging for the surgeon because Intraoperative Floppy Iris Syndrome (IFIS) might occur. However, the question is whether this has any practical implication for the outcomes of surgery. In this study we investigate whether cornea is damage during surgery on Tamsulosin patient. In an observational study 30 cataract patients taking Tamsulosin is compared to 30 patients not taking Tamsulosin, but otherwise similar. Number of patients is based on power calculation.

Cornea is examined by specular microscopy.

ELIGIBILITY:
Inclusion Criteria:

* cataract needing surgery

Exclusion Criteria:

* glaucoma
* corneal scarring
* diabetes
* uveitis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for catarct surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
corneal endothelium cell loss | 3 months
  Corneal endothelium cells was evaluated by specular microskopy before and 3 month post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Frederiksberg University Hospital, Frederiksberg, Frederiksberg, Denmark